CLINICAL TRIAL: NCT02216149
Title: Effects of S-1 and Capecitabine in Combination With Oxaliplatin on the Coronary Artery Blood Flow in Patients Metastatic Gastrointestinal Tract Adenocarcinoma: a Randomized Phase II Study
Brief Title: Effects of S-1 and Capecitabine on Coronary Artery Blood Flow
Acronym: FluoHeart
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Heikki Joensuu (Other)
Responsible Party: Sponsor-Investigator, Heikki Joensuu, MD, professor, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HUS-01/2013; 2013-003976-11 (EudraCT Number)
Record Dates: First submitted 2014-08-07; First posted 2014-08-13 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Esophagus Cancer; Stomach Cancer; Small Bowel Cancer; Colon Cancer; Rectum Cancer
Keywords: fluoropyrimidine; S-1; Teysuno; oxaliplatin; coronary artery flow; coronary artery dysfunction; gastrointestinal tract cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Gastrointestinal Neoplasms | interventions — S 1 (combination); tegafur-gimeracil-oteracil; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-1 plus oxaliplatin (SOX) (Experimental): Oxaliplatin 130 mg/m2 d. 1 followed by oral S-1 25 mg/m2/day BID d1-14.
  Interventions: Drug: S-1; Drug: Oxaliplatin
- Oxaliplatin plus capecitabine (XELOX) (Active Comparator): Intravenous oxaliplatin 130 mg/m2 d.1 followed by oral capecitabine 2000 mg/m2/day divided in 2 daily doses d1-14.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: S-1 — S-1 25 mg/m2/day BID d1-14, oxaliplatin injection 130 mg/m2 D1 every 3 weeks
  Other Names: Teysuno; tegafur/gimeracil/oteracil
  Arms: S-1 plus oxaliplatin (SOX)
Drug: Capecitabine — capecitabine 2000 mg/m2/day divided in 2 daily doses d1-14, oxaliplatin injection 130 mg/m2 D1 every 3 weeks
  Other Names: Xeloda
  Arms: Oxaliplatin plus capecitabine (XELOX)
Drug: Oxaliplatin — Oxaliplatin 130 mg/m2 D1 every 3 weeks
  Other Names: Eloxatin

SUMMARY:
Fluoropyrimidine chemotherapy agents , such as 5-fluorouracil and capecitabine, are occasionally associated with cardiac toxicity. Clinical fluoropyrimidine cardiotoxicity is infrequent, but subclinical toxicity may be much more common. Cardiac toxicity may be less frequent with S-1 as compared with 5-fluorouracil and capecitabine, but head-to-head comparisons are lacking. The purpose of the study is to compare 2 measures of subclinical coronary artery microvascular dysfunction, the coronary flow reserve and the coronary flow response to a cold pressor test, in a patient population who are being treated for adenocarcinoma of the gastrointestinal tract with one of 2 oxaliplatin-containing regimens, either with oxaliplatin plus S-1 or with oxaliplatin plus capecitabine.

DETAILED DESCRIPTION:
Patients diagnosed with adenocarcinoma of the gastroesophageal tract are randomly assigned to receive two 3-weekly cycles of either XELOX (intravenous oxaliplatin 130 mg/m2 d.1 followed by oral capecitabine 2000 mg/m2/day divided in 2 daily doses d1-14) or SOX (intravenous oxaliplatin 130 mg/m2 d. 1 followed by oral S-1 25 mg/m2/day BID d1-14). A cross-over between the 2 arms is carried out after the first 2 cycles; patients allocated to XELOX will receive 2 cycles of SOX (cycles 3 and 4), and those allocated to SOX will receive XELOX (cycles 3 and 4). Monitoring of the coronary artery flow, cardiac arrythmias, cardiac symptoms and blood biochemistry is done at baseline, during each chemotherapy cycle (cycles 1 to 4) and after treatment.Study treatment will continue until all patients have discontinued from treatment or maximum 24 weeks from the date of the first day of treatment, whichever occurs first. At that point, treatment may continue at the discretion of the Investigator. Each patient will be followed for survival status for a minimum of 12 months after first dose of study medication. Tumor assessments will be performed throughout the study period and analyzed using Response Evaluation Criteria in Solid Tumors (RECIST) criteria (Version 1.1, 2009). Computed tomography (CT) scans will be performed at the end of every 2 cycles. Cardiac assessments will be performed and analyzed using non-invasive transthoracic Doppler echocardiography, 24-h Holter registration, and plasma troponin concentration.

ELIGIBILITY:
Inclusion Criteria:

* Has given written informed consent.
* Is at least 18 years of age.
* Has advanced or metastatic gastrointestinal tract adenocarcinoma.
* No previous cancer chemotherapy for cancer.
* Measurable or evaluable lesions according to RECIST v1.1 criteria.
* Is able to take medications orally.
* Has ECOG performance status 0 or 1.
* Has a life expectancy of at least 3 months.
* Has adequate organ function.

Exclusion Criteria:

* Cancer considered operable without prior chemotherapy.
* Prior chemotherapy to cancer.
* Previous therapy with fluoropyrimidines or anthracyclines for any indication.
* Inability to swallow tablets.
* Known brain metastasis or leptomeningeal metastasis.
* History of myocardial infarction, coronary stenting/graft.
* History of unstable angina, coronary/peripheral artery bypass graft.
* History of cerebrovascular accident or transient ischemic attack.
* History of pulmonary embolism or deep vein thrombosis.
* Symptomatic congestive heart failure.
* Ongoing cardiac dysrhythmias.
* Patients with any cardiac disease that requires regular medication.
* Hypertensive crisis or severe hypertension that is not controlled.
* Is a pregnant or lactating female.
* The cardiac arterial flow tests cannot be done.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Frequency of coronary artery dysfunction | 3 months
  The frequency of subclinical coronary artery dysfunction is as assessed by comparing the coronary flow reserve during chemotherapy with the baseline coronary flow reserve, and the coronary flow response to a cold pressor test.

SECONDARY OUTCOMES:
Coronary artery blood flow rate | 3 months
  The coronary artery blood flow rate is measured with ultrasound. The rates are compared with the baseline and between the groups.
Cardiac arrythmias during 24-hour electrocardiogram registration | 3 months
  Cardiac arrythmias detected with Holter cardiac recording.
Adverse events between the allocation groups | 3 months
  by CTCAE.4
Response to chemotherapy | 3 months
  by RECIST 1.1
Survival status | 12 months
  Survival from the first dose of study medication to study completion

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Joensuu, MD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland